CLINICAL TRIAL: NCT07060950
Title: Analysis of Circulating Tumor Markers in Blood - ALCINA 5
Acronym: ALCINA 5
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROICM 2022-02 ALC
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Interventional study (blood collections and possibly tumor sample collection depending on cohort type) on single group cohorts (each cohort is defined in the arms below).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COHORT 1 - CURE (Other): Patients with histologically proven metastatic non-small cell lung carcinoma eligible for immunotherapy
  Interventions: Biological: Blood sampling C1

INTERVENTIONS:
Biological: Blood sampling C1 — Blood samples will be collected at four key time points :
  * baseline (T1),
  * first scan assessment (T2),
  * second scan assessment (T3),
  * and progression (T4).

SUMMARY:
The circulating tumoral biomarkers in the blood are the object of numerous researches for several decades. The potential clinical interests of these circulating biomarkers are diagnostic, prognostic, predictive of the efficiency of targeted therapies (according to the mutational profile of the cancer), and could allow the study of the mechanisms of resistance under process. In the multiplicity of these blood potential biomarkers joins a permanent evolution of the technological means used to detect them/to quantify, as well as to estimate their clinical utility.

DETAILED DESCRIPTION:
The new major challenge in research focuses on the rapid evaluation of circulating biomarker candidates, which could replace or complement molecular analyses of tumor tissue obtained through biopsy (for example the search for somatic mutations of cancer) by a simple blood test (liquid biopsy). The other current important challenge is to have an idea of the interest to analyse the kinetics of blood markers, in particular in answer to a clinical "event", either through the chemotherapy, a biopsy and / or surgery. There is almost no data in the literature on this aspect. It is very likely that the liberation in the blood of the blood tumoral markers is strongly dependent on medical interventions on the tumour.

The study ALCINA 5 relies exactly on the principle of small cohorts based on the analysis of circulating tumour biomarkers obtained by blood sampling, with comparison - if necessary - with tumour material obtained by biopsy. Which cohort correspond each to a clinical situation and/or a technique of different implemented detection. In case of success, statistical hypotheses will be necessary for the implementation of wider studies (being then the object of a specific approval by competent authorities).

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting an invasive tumoral pathology (proved or suspected), whatever is the location or the stage,
2. 18 years old or higher ?
3. Patient who has provided informed, written, and explicit consent,
4. Patient affiliated with a French Social Protection System.

   In the case of a tumor biopsy:
5. Tumor considered as accessible by biopsy,
6. Normal hemostasis assessment (PT, APTT, platelets),
7. No anticoagulant or antiaggregant treatment for the biopsy.

Exclusion Criteria:

1. Pregnant woman and/or breast-feeding,
2. Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons,
3. Private persons of freedom or under guardianship,
4. Patient with a history of other invasive cancers within the 5 years preceding inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
All Cohorts : Study of the feasibility of detecting and/or analysing blood or tissue tumour biomarkers. | 10 years
  Success rate of the detection technique used (the criterion will be detailed according to the biomarker evaluated, in each of the cohorts)

SECONDARY OUTCOMES:
COHORT 1 - CURE : to define a liquid biopsy signature for predicting therapeutic response from samples taken before initiation of immunotherapy (T1). | 4 years
  CTCs-PD-L1+/-, ctDNA, circulating proteins (CPs) and circulating immune cells (CICs) will be measured in accordance with the definitions established in T1.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France, France